CLINICAL TRIAL: NCT03165643
Title: Epigenetic Alteration of Rho Guanine Nucleotide Exchange Factor 11 (ARHGEF11) in Cord Blood Samples in Macrosomia Exposed to Intrauterine Hyperglycaemia
Brief Title: The DNA Methylation of ARHGEF11 in Macrosomia
Status: Completed | Type: Observational
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Jie Yan, Peking University First Hospital
Other Study IDs: 2013572
Record Dates: First submitted 2017-05-21; First posted 2017-05-24 (Actual); Last update posted 2017-05-24 (Actual); Status verified 2017-05

CONDITIONS: Gestational Diabetes; Diabetes; Macrosomia, Fetal
MeSH Terms: conditions — Diabetes, Gestational; Diabetes Mellitus; Fetal Macrosomia | interventions — Glucose Tolerance Test

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- NGT-normal birth weight
- NGT-macrosomia
- GDM-normal birth weight
  Interventions: Diagnostic Test: OGTT
- GDM-macrosomia
  Interventions: Diagnostic Test: OGTT

INTERVENTIONS:
Diagnostic Test: OGTT — 75 g glucose tolerance test was provided to all pregnant women during 24-28 weeks.
  Groups: GDM-macrosomia; GDM-normal birth weight

SUMMARY:
Background Macrosomia at birth is associated with subsequent susceptibility to obesity, abnormal glucose metabolism, hypertension and dyslipidaemia. Epigenetic reprogramming has been reported to be involved in the development of human diseases caused by suboptimal environmental or nutritional factors.

Objective The study was aiming to explore epigenetic mechanism influences on macrosomic infants exposed to intrauterine hyperglycemia.

Design The investigators performed a genome-wide analysis of DNA methylation in cord blood from macrosomic infants born to women with gestational diabetes or infants with normal birth weight born to normal glucose-tolerant women in order to identify genes related to foetal growth or early adipose tissue development. The candidate genes were then validated using SEQUENOM MassARRAY after bisulfite conversion.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* Pregnancies complicating with hypertensive disorders, pre-gestational diabetes, thyroid diseases, renal dysfunction were excluded.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Singleton term pregnant women in Peking University First Hospital were recruited in this study.
Sampling Method: Non-Probability Sample
Enrollment: 239 (Actual)
Dates: Start 2014-03-06 (Actual); Primary Completion 2014-10-18 (Actual); Study Completion 2014-10-18 (Actual)

PRIMARY OUTCOMES:
GDM was identified | 24-28 weeks
  According to the International Association of Diabetes and Pregnancy Study Groups (IADPSG) criteria, gestational diabetes mellitus (GDM) was diagnosed when at least one cut point was reached in 2-hour 75-g OGTT test: a fasting plasma glucose (FPG) ≥ 5.1 mmol/L (92 mg/dL), a 1-hour ≥ 10.0 mmol/L (180 mg/dL) or a 2-hour ≥ 8.5 mmol/L (153 mg/dL). Participants were divided into two groups based on OGTT: Group normal glucose tolerant (NGT, n=132) and Group GDM (n=107).
Foetal macrosomia was identified | 40 weeks
  After delivery, participants were further divided into four subgroups based on neonatal birth weight: normal birth weight (NBW) was defined as 2500g ≤ birth weight < 4000g, macrosomia (Mac) was defined as birth weight ≥ 4000g. Group NGT-NBW (n=83): normal glucose tolerant women with normal neonatal birth weight; Group NGT-Mac (n=49): normal glucose tolerant women with macrosomia; Group GDM-NBW (n=82): GDM women with normal neonatal birth weight; Group GDM-Mac (n=25): GDM women with macrosomia.
DNA methylation level in macrosomia | 40 weeks
  Investigators performed a genome-wide analysis of DNA methylation in cord blood from macrosomic infants born to women with gestational diabetes or infants with normal birth weight born to normal glucose-tolerant women in order to identify genes related to foetal growth or early adipose tissue development. The candidate genes were then validated using SEQUENOM MassARRAY after bisulfite conversion.